CLINICAL TRIAL: NCT06650566
Title: A Phase I/II, Open-label, Dose Escalation and Dose Expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of LM-299 Injection as Monotherapy or in Combination With Other Anti-tumor Therapies in Patients With Advanced Solid Tumors
Brief Title: Study of LM-299 in Subjects Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM299-01-102
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-11

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-299 Dose Escalation at different dose levels (Experimental)
  Interventions: Drug: LM-299
- LM-299 Dose Escalation Backfill Cohorts (Experimental)
  Interventions: Drug: LM-299

INTERVENTIONS:
Drug: LM-299 — Q2W/Q3W,Intravenous Drip

SUMMARY:
For Phase I Dose Escalation Stage, to assess the safety and tolerability of LM-299 in patients with advanced solid tumors,determine the maximum tolerated dose (MTD) or optimal biological dose (OBD), and explorethe recommended dose for expansion (RDE) in patients with advanced solid tumours..

For Phase II Dose Expansion Stage, to assess the antitumor activity of LM-299 in patients with various advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Participant must be 18- 18 years or the legal age of consent at the time of signing the ICF.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Life expectancy ≥ 3 months.
5. Patients with advanced solid tumors confirmed by histopathological diagnosis who have failed standard treatment, are intolerant to standard treatment, or for whom standard treatment is currently unsuitable.
6. Pre-treatment archived tumour tissue (within 5 years) or fresh samples could be provided for biomarker analysis.
7. Must have at least one measurable lesion according to RECIST v1.1.
8. Adequate organ and bone marrow function as defined by protocol.
9. Female subjects of childbearing potential or male subjects with partners of childbearing potential agree to use highly effective contraception.
10. Subjects who are able to communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Participate in any other clinical trial within 28 days prior to 1st dosing of LM-299.
2. Subjects who have received the anti-tumor treatments within the specified time periods prior to the first dosing of LM-299.
3. Any adverse event from prior anti-tumour therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
4. Subjects with uncontrolled tumour-related pain.
5. Subjects with known central nervous system (CNS) or meningeal metastasis.
6. Qualitative urine protein results ≥ 3+.
7. Clinically significant hemoptysis or tumor bleeding within 2 weeks prior to 1st dosing of LM-299.
8. Any life-threatening bleeding event that occurred within 3 months prior to 1st dosing of LM-299.
9. Subjects with esophageal or gastric varices requiring immediate intervention or a history of variceal bleeding .
10. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh class B or more severe liver cirrhosis.
11. Subjects who have clinically uncontrollable third-space fluid accumulatio.
12. Radiographic evidence of tumor invading surrounding vital organs or the risk of esophagotracheal fistula or esophagopleural fistula, tumor surrounding or invading the major blood vessels, or presence of intratumoral cavity formation.
13. History of gastrointestinal perforation and/or fistula within 6 months prior to the first dose of the study drug.
14. Patients with complete or incomplete intestinal obstruction within 3 months prior to the first dose of the study drug or patientswho are currently at the risk of intestinal perforation.
15. Subjects who are known to be allergic to antibody treatment.
16. Subjects who take systemic corticosteroids (≥ 10 mg/day of prednisone or equivalent) for more than 7 days within 2 weeks prior to the first dose of LM-299.
17. Subjects with the known history of autoimmune disease.
18. Patients with a history of active or previously confirmed inflammatory bowel disease.
19. Patients with a history of or currently having interstitial pneumonia requiring systemic corticosteroid treatment.
20. Received live vaccines or attenuated live vaccines within 28 days prior to the first dose of the study drug.
21. Currently using anticoagulants such as therapeutic doses of heparin or vitamin K antagonists.
22. Subjects who received major surgery or interventional treatment within 28 days prior to 1st dosing of LM-299 (excluding tumour biopsy, puncture, etc.).
23. Subjects who have severe cardiovascular and and cerebrovascular diseases.
24. Patients with severe infections within 4 weeks prior to the first dose.
25. Patients with a history of immunodeficiency.
26. Individuals with HIV infection, active HBV or HCV infection .
27. Patients with known active tuberculosis (TB). Suspected active TB should be ruled out through clinical examination.
28. Patients who have had other malignancies within 5 years prior to the first dose of the study drug.
29. Women of childbearing age who test positive for pregnancy within 7 days prior to the first dose of the study drug or are breastfeeding.
30. Individuals with known psychiatric disorders or illnesses that may affect adherence to the trial.
31. Patients with local or systemic diseases caused by non-malignant tumors.
32. Subject who is judged as not eligible to participate in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limitingtoxicity (DLT) | 53 weeks
  Phase 1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 53 weeks
  Phase 1
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | 53 weeks
  Phase 1
Overall Response Rate (ORR) | 50 weeks
  Phase 2

SECONDARY OUTCOMES:
PK Parameter: Area Under the Concentration-time Curve(AUClast) | 103 weeks
  Phase 1 and 2
PK Parameter: Area Under the Concentration-time Curve(AUCtau) | 103 weeks
  Phase 1 and 2
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) | 103 weeks
  Phase 1 and 2
PK Parameter:Time of Maximum Observed Concentration (Tmax) | 103 weeks
  Phase 1 and 2
PK Parameter: Elimination Half-life (t1/2) | 103 weeks
  Phase 1 and 2
PK Parameter: Steady State Maximum Concentration(Cmax,ss) | 103 weeks
  Phase 1 and 2
PK Parameter: Steady State Minimum Concentration(Cmin,ss) | 103 weeks
  Phase 1 and 2
PK Parameter: Systemic Clearance at Steady State (CLss) | 103 weeks
  Phase 1 and 2
PK Parameter: Volume of Distribution at Steady-State (Vss) | 103 weeks
  Phase 1 and 2
PK Parameter: Accumulation Ratio (Rac AUC) | 103 weeks
  Phase 1 and 2
PK Parameter: Degree of Fluctuation (DF) | 103 weeks
  Phase 1 and 2
Overall Response Rate (ORR) | 53 weeks
  Phase 1
Duration of Response (DOR) in Month | 103 weeks
  Phase 1 and 2
Disease control rate (DCR) in percentage | 103 weeks
  Phase 1 and 2
progression-free survival (PFS) in Month | 103 weeks
  Phase 1 and 2
Overall survival (OS) in Month | 103 weeks
  Phase 1 and 2
PK Parameter: Accumulation Ratio (Rac Cmax) | 103 weeks
  Phase 1 and 2

CONTACTS AND LOCATIONS:
Locations (6):
- One Clinical Research, Perth, Western Australia, Australia
- China (5):
  - the first affiliated hospital of Xinxiang medical University, Xinxiang, Henan
  - Liaocheng people's hospital, Liaocheng, Shandong
  - Zibo municipal hospital, Zibo, Shandong
  - Shanghai Dongfang Hospital (Tongji University Affiliated Dongfang Hospital), Shanghai, Shanghai Municipality
  - Shanghai GoBroad Cancer Hospital China Pharmaceutical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No